CLINICAL TRIAL: NCT04220346
Title: The Effect of Playing Games With Tablet on Pain and Anxiety During Circumcision in Children: A Randomized Controlled Study
Brief Title: Distraction Method on Pain and Anxiety During Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-123
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Pain; Anxiety; Urological Nursing
Keywords: anxiety; children; circumcision; nursing; pain
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet group (Experimental): The Tablet group played the game with Tablet during the whole circumcision.
  Interventions: Other: Tablet group
- Control group (No Intervention): The control group did not play game with Tablet during the procedure.

INTERVENTIONS:
Other: Tablet group — Children in the Tablet group started to play the game with Tablet about 5-10 minutes before circumcision, and continued to play the game during the whole procedure.
  Arms: Tablet group

SUMMARY:
Circumcision is a common procedure in infants, children and young people around the world for cultural, religious or medical reasons. Since this is a painful procedure, it is performed under local anesthesia or general anesthesia. It is recommended to perform this procedure under local anesthesia if there is no risk. Although local anesthesia is used during the procedure, pain and anxiety levels of children may increase. Distraction methods are commonly used and effective methods to reduce pain and anxiety during painful procedures. The aim of this study was to evaluate the effect of tablet playing during circumcision on pain and anxiety in school age children.

DETAILED DESCRIPTION:
Circumcision is a common procedure in the worldwide. To our knowledge, although there have been several randomized controlled trials using video and game techniques, which are distractions to reduce pain and anxiety during painful procedures, no randomized controlled trials using playing the game with Tablet to reduce pain and anxiety during circumcision have been found. Non-pharmacological studies, such as play therapy, are needed to reduce pain and anxiety in school-age children undergoing circumcision under local anesthesia. The aim of this study is to provide evidence about the effectiveness of playing the game with Tablet used to reduce pain and anxiety during circumcision, and to contribute to nursing care in pain management.

ELIGIBILITY:
Inclusion Criteria:

* being between 7-12 years
* male gender
* circumcision with local anesthesia
* agreeing to participate in the study

Exclusion Criteria:

* presence of any contraindication for circumcision (hemophilia, bleeding disorders, urinary anatomical disorders-hypospadias, epispadias etc.)
* any analgesic used 24 hours before circumcision

Ages: 7 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
change on pain intensity as measured by Visual Analog Scale | "5-10 minutes before procedure", "during procedure" and "5 minutes after" circumcision.
  The average score change on pain intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure pain intensity. The scale is a measuring tool with length of 0-10 cm (0-100 mm). High scores on the scale indicate that pain intensity is high.

SECONDARY OUTCOMES:
score change on anxiety level as measured by State-Trait Anxiety Inventory for Children | "5-10 minutes before procedure" and "5 minutes after procedure" circumcision.
  The average score change on anxiety level as measured by State-Trait Anxiety Inventory for Children. This scale is used to measure anxiety. The scores on the scale ranges from 20 to 60. The high scores on the scale indicate that anxiety is high.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, RN, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussein HA. Effect of active and passive distraction on decreasing pain associated with painful medical procedures among school aged children. World Journal of Nursing Sciences 1(2): 13-23, 2015.
- [Background] Liguori S, Stacchini M, Ciofi D, Olivini N, Bisogni S, Festini F. Effectiveness of an App for Reducing Preoperative Anxiety in Children: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):e160533. doi: 10.1001/jamapediatrics.2016.0533. Epub 2016 Aug 1. PMID 27294708
- [Background] Polat F, Tuncel A, Balci M, Aslan Y, Sacan O, Kisa C, Kayali M, Atan A. Comparison of local anesthetic effects of lidocaine versus tramadol and effect of child anxiety on pain level in circumcision procedure. J Pediatr Urol. 2013 Oct;9(5):670-4. doi: 10.1016/j.jpurol.2012.07.022. Epub 2012 Sep 7. PMID 22959557
- [Background] Rizalar S, Tural Buyuk E, Yildirim N. Children's perspectives on the medical and cultural aspects of circumcision. Iranian Journal of Pediatrics 27(2): 1-7, 2017.
- [Background] Wilson-Smith EM. Procedural Pain Management in Neonates, Infants and Children. Rev Pain. 2011 Sep;5(3):4-12. doi: 10.1177/204946371100500303. PMID 26526331
- [Background] American Academy of Pediatrics Task Force on Circumcision. Circumcision policy statement. Pediatrics. 2012 Sep;130(3):585-6. doi: 10.1542/peds.2012-1989. Epub 2012 Aug 27. PMID 22926180